CLINICAL TRIAL: NCT05721534
Title: Effective Deprescribing in Primary Care Without Deterioration of Health-related Outcomes
Brief Title: Deprescribing and Health-related Effects
Status: Completed | Type: Observational
Sponsor: Anne Estrup Olesen (Other)
Collaborators: Frederikshavn Kommune, Frederikshavn, Denmark (Unknown); Lægeklinikken Frederikshavn, Frederikshavn, Denmark (Unknown)
Responsible Party: Sponsor-Investigator, Anne Estrup Olesen, Professor, Aalborg University Hospital
Organization: Aalborg University Hospital (Other)
Other Study IDs: K2023-008
Record Dates: First submitted 2023-02-01; First posted 2023-02-10 (Actual); Last update posted 2023-02-10 (Actual); Status verified 2023-02

CONDITIONS: Chronic Disease
Keywords: Primary care; Medication review; Deprescribing; Polypharmacy; Chronic disease management
MeSH Terms: conditions — Chronic Disease | interventions — Medication Review

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Care home residents: The intervention was offered to new residents and residents that had not yet attended a consultation focusing on pharmacological treatment in The Chronic Care Model.
  Interventions: Other: Medication review
- Community-dwelling patients with chronic disease: Patients were invited for the consultation focusing on pharmacological treatment in the month of their birthday and, thereby, included randomly and consecutively throughout the study period.
  Interventions: Other: Medication review

INTERVENTIONS:
Other: Medication review — Annual consultation focusing on pharmacological treatment. This specific consultation constituted the "intervention". It included a structured review of the patient's health state, in addition to a structured medication review with a focus on appropriate medication and deprescribing.
  Other Names: Medication review with focus on deprescribing

SUMMARY:
In a primary care settled quality improvement project aiming to deprescribe medication through a medication review intervention, we investigated how the implemented medication changes affected health-related outcomes in real-life patients.

DETAILED DESCRIPTION:
The project was approved by the Management in the Municipality of Frederikshavn. According to Danish legislation, no formal permission from the national or regional Committee on Health Research Ethics was required for this type of study, as patients were not treated inferior to usual care and no biological material was collected. It was conducted as a quality improvement project and informed consent was not required for the specific data collected. The study is in compliance with the General Data Protection Regulation and a part of North Denmark Region's record of processing activities (K2023-008).

ELIGIBILITY:
Inclusion Criteria:

* new residents and residents that had not yet attended a consultation focusing on pharmacological treatment in The Chronic Care Model.
* patients were invited for the consultation focusing on pharmacological treatment in the month of their birthday and, thereby, included randomly and consecutively throughout the study period.

Exclusion Criteria:

* unable to collaborate on follow-up questionnaires

Ages: 50 Years to 105 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study included care home residents living in selected care homes, in which the GPF was associated "care home doctors", and community-dwelling patients with chronic disease listed with the GPF.
Sampling Method: Probability Sample
Enrollment: 87 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
self-reported health status | 4 months
  (on a scale from 1 to 10)

SECONDARY OUTCOMES:
general condition | 4 months
  (rated on a 5-point Likert Scale)
functional level | 4 months
  rated on a 5-point Likert Scale

CONTACTS AND LOCATIONS:
Overall Officials: Anne E Olesen, Study Chair — Professor
Locations (1):
- Aalborg University Hospital, Aalborg, Denmark

IPD SHARING:
Plan to Share IPD: No